CLINICAL TRIAL: NCT05847764
Title: Disitamab Vedotin Combined Therapy for Locally Advanced or Metastatic NSCLC With HER2 Alterations, a Phase II Study
Brief Title: Disitamab Vedotin Combined Therapy for Locally Advanced or Metastatic NSCLC Patients With HER2 Alterations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Head of Oncology Department, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCVDODIIR006
Record Dates: First submitted 2023-03-21; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Non Small Cell Lung Cancer; ERBB2 Mutation-Related Tumors; RC48; Disitamab Vedotin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: RC48+PD-1/PD-L1 inhibitor (Experimental)
  Interventions: Drug: RC48+Tislelizumab+carboplatin
- Arm 2: RC48+Furmonertinib, 1L (Experimental)
  Interventions: Drug: RC48+Furmonertinib, 1L
- Arm 3: RC48+Furmonertinib, 2L+ (Experimental)
  Interventions: Drug: RC48+Furmonertinib, 2L+

INTERVENTIONS:
Drug: RC48+Tislelizumab+carboplatin — RC48+PD-1/PD-L1 inhibitor+chemo in treatment-naive patients harboring HER2 alterations
  Arms: Arm 1: RC48+PD-1/PD-L1 inhibitor
Drug: RC48+Furmonertinib, 1L — RC48+Furmonertinib in treatment-naive patients harboring EGFR mutations as well as HER2 alterations
  Arms: Arm 2: RC48+Furmonertinib, 1L
Drug: RC48+Furmonertinib, 2L+ — RC48+Furmonertinib in patients who failed at least one line of standard treatment and harboring HER2 alterations
  Arms: Arm 3: RC48+Furmonertinib, 2L+

SUMMARY:
Disitamab Vedotin combined therapy locally advanced or metastatic NSCLC Patients with HER2 Alterations.

DETAILED DESCRIPTION:
This study will explore the treatment of locally advanced or metastatic non-small cell lung cancer with HER2 mutation, amplification, or HER2 mutation (mutation, amplification, protein over-expression) using Disitamab Vedotin（RC48） combined with Tislelizumab or third-generation EGFR-TKI Furmonertinib, in the aim of providing new treatment strategies for lung cancer patients with HER2 pathway activation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 (inclusive) or above, regardless of gender.
2. Histologically or cytologically confirmed locally advanced or metastatic NSCLC, not suitable for radical surgery or radiotherapy (TNM 8th Edition).".
3. Biomarker:

   * Arm 1: HER2 alterations, no other driver gene mutations；
   * Arm 2: EGFR mutations accompanied by HER2 alterations;
   * Arm 3: HER2 gene mutations, no other driver gene alterations;
4. Number of treatment lines:

   * Arm 1-2: patients who have not previously received systemic treatment for advanced diseases;
   * Arm3:Failed with at least one line of standard treatment or intolerance;
5. Patients who have previously undergone neoadjuvant chemotherapy, adjuvant chemotherapy, radiotherapy, or radiochemotherapy for the purpose of curing non metastatic diseases must have a disease-free interval of 6 months from the last chemotherapy and/or radiotherapy to the randomization date.
6. There is at least one measurable lesion that meets the definition of the RECIST 1.1 standard at baseline.
7. ECOG fitness status score: 0 or 1 point.
8. Estimated survival time ≥ 3 months.

Exclusion Criteria:

1. Central nervous system metastasis or meningeal metastasis with clinical symptoms.
2. Have a history of autoimmune diseases, immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
3. Active hepatitis B (hepatitis B virus titer>1000 copies/ml or 200 IU/ml); Hepatitis C virus and syphilis infection.
4. Have undergone major organ surgery (excluding puncture biopsy) or have experienced significant trauma within 3 weeks before the first use of the study drug.
5. Known hypersensitivity or intolerance to any component of the study protocol drug or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Objective Response Rate (ORR) Based on Investigator Assessment Following Treatment in Participants With HER2 alterations Non-Small-Cell Lung Cancer (NSCLC) | Up to 24 months (data cut-off)
  Percentage of Participants who have a complete response (CR) or partial response (PR) as assessed by investigator according to RECIST 1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) Following Treatment in Participants With HER2 alterations Non-Small-Cell Lung Cancer (NSCLC) | Up to 24 months (data cut-off)
  Defined as the proportion of participants who have a complete response (CR), partial response (PR) or standard disease (SD) as assessed by investigator according to RECIST 1.1
Progression-free survival (PFS) Following Treatment in Participants With HER2 alterations Non-Small-Cell Lung Cancer (NSCLC) | Up to 24 months (data cut-off)
  Defined as time from randomization until progression per RECIST 1.1 as assessed by investigator, or death due to any cause.
Duration of Response (DoR) Following Treatment in Participants With HER2 alterations Non-Small-Cell Lung Cancer (NSCLC) | Up to 24 months (data cut-off)
  Defined as the time from the date of first documented response until date of documented progression as assessed by investigator assessment according to RECIST 1.1.
Overall Survival (OS) Following Treatment in Participants With HER2 alterations Non-Small-Cell Lung Cancer (NSCLC) | Up to 24 months (data cut-off)
  Defined as time from randomization until the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Li PI Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- SunYat-senU, Guanzhou, China

IPD SHARING:
Plan to Share IPD: No